CLINICAL TRIAL: NCT01729897
Title: A Multicenter Open-label Randomized Controlled Clinical Trial of Etomidate Emulsion for Sedation in Patients Scheduled for Upper GI Endoscopy
Brief Title: Etomidate Emulsion for Sedation in Patients Scheduled for Upper Gastrointestinal (GI) Endoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jiangsu Nhwa Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChiCTR-TRC-20121001
Record Dates: First submitted 2012-10-18; First posted 2012-11-20 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: Complication of Gastrostomy
Keywords: gastroscopy; sedation; etomidate
MeSH Terms: interventions — Etomidate; Fentanyl; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Etomidate & Fentanyl (Experimental): * 4 min before procedure: fentanyl 1 μg/kg (0.02 ml/kg), intravenous injection
  * After injection of fentanyl, etomidate was infused intravenously at rate of 200 ml/h for 30 seconds with unified injection pump, then after interval time of 30 seconds, infusion rate was altered to 500 ml/h and infusion was sustained until patients fell asleep.
  * Additional dose of etomidate would be administrated separately when duration of procedure was prolonged.
  Interventions: Drug: Etomidate; Drug: Fentanyl
- Propofol & Fentanyl (Placebo Comparator): * 4 min before procedure: fentanyl 1 g/kg (0.02 ml/kg), intravenous injection
  * After injection of fentanyl, propofol was infused intravenously at rate of 200 ml/h for 30 seconds with unified injection pump, then after interval time of 30 seconds, infusion rate was altered to 500 ml/h and infusion was sustained until patients fell asleep.
  * Additional dose of propofol would be administrated separately when duration of procedure was prolonged.
  Interventions: Drug: Fentanyl; Drug: Propofol

INTERVENTIONS:
Drug: Etomidate
  Arms: Etomidate & Fentanyl
Drug: Fentanyl
Drug: Propofol
  Arms: Propofol & Fentanyl

SUMMARY:
The study is designed to explore and compare the efficacy and safety of etomidate and propofol with or without analgesic for painless gastroscopy, and to provide more reliant support for implementation and promotion of comfort care.

DETAILED DESCRIPTION:
To widely implement painless gastroscopy is required by diagnose and treatment with gastroscopy due to the large number and significant suffering of the patients. Also, development and exploration of anesthesiology will be bound to prompt the development and exploration of painless gastroscopy. However, the anesthesia risk of painless gastroscopy are usually higher than that of general anesthesia performed in operating room due to the condition, monitoring and equipments as well as the staffing for its implementation. Thus, the finding of a safe and convenient approach for general anesthesia will have a profound impact on a full promotion and implementation of comfortable care.

Etomidate, with the main advantage of little effect on circulatory and respiratory systems, and the features of rapid onset and metabolism, may be helpful to guarantee the safety of painless diagnosis and treatment, thus appropriate for the procedure with short duration of anesthesia. However, there is controversy regarding whether analgesic should be used in combination, as well as how to given the combined regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for painless gastroscopy
* 18-80 year old
* 18 H2 ≤ weight ≤ 35 H2 (H indicates height)
* American Society of Anesthesiologists (ASA) physical status class 1-3
* The duration of surgery is ≤ 60 min ( duration of surgery was defined as the interval time from insert to withdraw of catheter)
* Without liver, kidney and heart disease history
* No previous history of abnormal recovery of anesthesia in surgery

Exclusion Criteria:

* Patients whom do not wish to perform painless gastroscopy or participate in the study
* Patients with medical history of severe heart, lung, liver, kidney or metabolic disease
* Patients with abnormal ECG presented as heart rate 50 < beat/min
* Patients who suffered from acute inflammation of respiratory tract within the past 2 weeks and did not be cured of it before participating in the study
* Hypertension patient with preoperative blood pressure > 180/90 mmHg; hypotension patients with preoperative blood pressure < 90/60 mmHg;
* Patients with neuromuscular disease, mental disorders
* Hemoglobin is less than 90 g/L
* Patients with suspected abuse of Anesthesia and Analgesia
* Patients who were predicted to have or had previous difficult airway ( difficult airway is defined as the clinical situation in which a conventionally trained anesthesiologist experiences three failures of intubation)
* Patients with known emulsion or opioid allergy
* Patients who will be noncompliant or unable to communicate
* Patients who received long-term treatment with hormone or had history of adrenocortical suppression
* Patients received coadministration of other sedative, analgesic ( including injection, oral or usage of relevant Chinese patent medicine) before, during or 15 min after the procedure
* Patients who appeared nausea and vomit, dizziness
* Patients with sever diabetes mellitus, hyperkaliemia or significant electrolyte disturbances

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2012-05; Primary Completion 2012-08 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
the minimum blood pressure | participants will be followed for the duration that from the beginning of the surgery to the extraction of the gastroscopy, an expected average of 2 hours
the proportion of hypotension | participants will be followed for the duration that from the beginning of the surgery to the extraction of the gastroscopy, an expected average of 2 hours
the minimum oxygen saturation of blood | participants will be followed for the duration that from the beginning of the surgery to the extraction of the gastroscopy, an expected average of 2 hours
Time interval | from the last administration of etomidate to when the patient leave the hospital
  the time interval that from the last administration of etomidate to when the patient leave the hospital

SECONDARY OUTCOMES:
Incidence rate of the side effects | participants will be followed for the duration from the beginning of the surgery to leaving hospital，an expected average of 4 hours
  the side effects include dizziness，nausea，vomit，myoclonia，injection pain，and the awareness during operation
the cost of the experiment drug | the money that the participants spend from the beginning of the surgery to leaving hospital，an expected average of 4 hours

OTHER OUTCOMES:
Other adverse events except above | participants will be followed for the duration from the beginning of the surgery to leaving hospital，an expected average of 4 hours
the changes of the primary clinical symptoms | participants will be followed for the duration from the beginning of the surgery to leaving hospital，an expected average of 4 hours
the abnormal laboratory examinations | participants will be followed for the duration from the beginning of the surgery to leaving hospital，an expected average of 4 hours